CLINICAL TRIAL: NCT00033631
Title: A Phase III Randomized Study Of High Dose 3D-CRT/IMRT Versus Standard Dose 3D-CRT/IMRT In Patients Treated For Localized Prostate Cancer
Brief Title: Radiation Therapy in Treating Patients With Stage II Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0126; CDR0000069306
Record Dates: First submitted 2002-04-09; First posted 2003-01-27 (Estimated); Results first posted 2017-02-08 (Estimated); Last update posted 2023-01-18 (Actual); Status verified 2022-12

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IIB prostate cancer; stage IIA prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 70.2 Gy (Active Comparator): 70.2 Gy 3D-CRT/IMRT
  Interventions: Radiation: 70.2 Gy 3D-CRT/IMRT
- 79.2 Gy (Experimental): 79.2 Gy 3D-CRT/IMRT
  Interventions: Radiation: 79.2 Gy 3D-CRT/IMRT

INTERVENTIONS:
Radiation: 70.2 Gy 3D-CRT/IMRT — Radiation will be delivered via 3D conformal radiation therapy (3D-CRT) or intensity modulated radiation therapy (IMRT) in 1.8 Gy minimum dose fractions to a total of 70.2 Gy in 39 Fractions. All fields treated once daily, five fractions per week. No more than 2% of the planning target volume and none of the clinical target volume may receive less than 70.2 Gy.
  Other Names: 3D conformal radiation therapy; intensity modulated radiation therapy
  Arms: 70.2 Gy
Radiation: 79.2 Gy 3D-CRT/IMRT — Radiation will be delivered via 3D conformal radiation therapy (3D-CRT) or intensity modulated radiation therapy (IMRT) in 1.8 Gy minimum dose fractions to a total of 79.2 Gy in 44 fractions. All fields treated once daily, five fractions per week. No more than 2% of the planning target volume and none of the clinical target volume may receive less than 79.2 Gy.
  Other Names: 3D conformal radiation therapy; intensity modulated radiation therapy
  Arms: 79.2 Gy

SUMMARY:
RATIONALE: Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. It is not yet known which dose of radiation therapy is more effective in treating stage II prostate cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of two different doses of specialized radiation therapy in treating patients who have stage II prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival of patients with stage II adenocarcinoma of the prostate treated with high- vs standard-dose three-dimensional conformal or intensity-modulated radiotherapy.
* Compare the freedom from prostate-specific antigen failure, disease-specific survival, local progression, and distant metastases in patients treated with these regimens.
* Compare the probability of tumor control and normal tissue complications in patients treated with these regimens.
* Compare the incidence of grade 2 or greater genitourinary and gastrointestinal acute and late toxicity in patients treated with these regimens.
* Compare the quality of life, including sexual function, of patients treated with these regimens.
* Correlate histopathologic or tumor-specific cytogenetic or chromosomal markers with cancer control outcomes in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to Gleason score and prostate-specific antigen (PSA) level (Gleason score 2-6, PSA ≥10 mg/mL but < 20 ng/mL vs Gleason score 7, PSA < 15 ng/mL) and radiation modality (three-dimensional conformal radiotherapy [3D-CRT] vs intensity-modulated radiotherapy [IMRT]). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo standard-dose 3D-CRT or IMRT once daily, 5 days a week, for 7.8 weeks (39 treatment days).
* Arm II: Patients undergo high-dose 3D-CRT or IMRT once daily, 5 days a week, for 8.8 weeks (44 treatment days).

Quality of life (QOL) is assessed initially at baseline. After completion of radiotherapy, QOL is assessed every 3 months for 1 year and then every 6 months for 4 years.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 1,520 patients (760 per treatment arm) will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Clinical stage T1b-T2b
* Meets one of the following criteria:

  * Gleason score 2-6 AND prostate-specific antigen (PSA) ≥ 10 ng/mL but < 20 ng/mL
  * Gleason score 7 AND PSA < 15 ng/mL
* No regional lymph node involvement
* No distant metastases

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* Zubrod 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No other invasive malignancy within the past 5 years except localized basal cell or squamous cell skin cancer
* No other major medical or psychiatric illness that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior cytotoxic chemotherapy
* No concurrent cytotoxic chemotherapy

Endocrine therapy:

* At least 3 months since prior finasteride
* No other prior hormonal therapy, including:

  * Luteinizing hormone-releasing hormone agonists (e.g., goserelin or leuprolide)
  * Antiandrogens (e.g., flutamide or bicalutamide)
  * Estrogens (e.g., diethylstilbestrol)
* No concurrent (neoadjuvant or adjuvant) hormonal therapy

Radiotherapy:

* No prior pelvic irradiation or brachytherapy

Surgery:

* No prior radical surgery (prostatectomy) or cryosurgery for prostate cancer
* No prior surgical castration (bilateral orchiectomy)

Other:

* At least 3 months since prior finasteride or phytoestrogen preparation (PC-SPES)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1534 (Actual)
Dates: Start 2002-03; Primary Completion 2014-04 (Actual); Study Completion 2022-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff M. Michalski, MD, Principal Investigator — Washington University - Saint Louis; James Purdy, Ph.D., Study Chair — UC Davis; Deborah W Bruner, Ph.D., Study Chair — Emory University; Mahul Amin, M.D., Study Chair — Cedars-Sinai
Locations (86):
- United States (72):
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - Radiological Associates of Sacramento Medical Group, Incorporated, Sacramento, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Washington Cancer Institute at Washington Hospital Center, Washington D.C., District of Columbia
  - Bay Medical, Panama City, Florida
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Oncology Center at Saint Margaret Mercy Healthcare Center, Hammond, Indiana
  - Cancer Center at Ball Memorial Hospital, Muncie, Indiana
  - Providence Medical Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Johnson County Radiation Therapy, Overland Park, Kansas
  - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Central Maryland Oncology Center, Columbia, Maryland
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Independence Regional Health Center, Independence, Missouri
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - Kansas City Cancer Center at St. Joseph's Medical Mall, Kansas City, Missouri
  - St. Joseph Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Parvin Radiation Oncology, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Radiation Oncology Associates of Kansas City at Northland Radiation Oncology Center, Kansas City, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Cancer Institute of New Jersey at Cooper University Hospital - Camden, Camden, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Lovelace Medical Center - Downtown, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - New York Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Cancer Centers of North Carolina - Raleigh, Raleigh, North Carolina
  - Rex Cancer Center at Rex Hospital, Raleigh, North Carolina
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Precision Radiotherapy at University Pointe, West Chester, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - MNAP Oncologic Center, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - CCOP - Main Line Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Danville Regional Medical Center, Danville, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Community Memorial Hospital Cancer Care Center, Menomonee Falls, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - All Saints Cancer Center at Wheaton Franciscan Healthcare, Racine, Wisconsin
- Canada (14):
  - Tom Baker Cancer Centre - Calgary, Calgary, Alberta
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Doctor H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - Northeastern Ontario Regional Cancer Centre, Greater Sudbury, Ontario
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Cancer Care Program at Thunder Bay Regional Health Sciences, Thunder Bay, Ontario
  - Edmond Odette Cancer Centre at Sunnybrook, Toronto, Ontario
  - Hopital Notre-Dame du CHUM, Montreal, Quebec
  - McGill Cancer Centre at McGill University, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan

REFERENCES:
- [Background] Cranmer-Sargison G. A treatment planning investigation into the dosimetric effects of systematic prostate patient rotational set-up errors. Med Dosim. 2008 Autumn;33(3):199-205. doi: 10.1016/j.meddos.2007.06.005. PMID 18674684
- [Result] Potrebko PS, McCurdy BM, Butler JB, El-Gubtan AS, Nugent Z. Optimal starting gantry angles using equiangular-spaced beams with intensity modulated radiation therapy for prostate cancer on RTOG 0126: a clinical study of 5 and 7 fields. Radiother Oncol. 2007 Nov;85(2):299-305. doi: 10.1016/j.radonc.2007.06.019. Epub 2007 Sep 7. PMID 17825932
- [Derived] Spratt DE, Tang S, Sun Y, Huang HC, Chen E, Mohamad O, Armstrong AJ, Tward JD, Nguyen PL, Lang JM, Zhang J, Mitani A, Simko JP, DeVries S, van der Wal D, Pinckaers H, Monson JM, Campbell HA, Wallace J, Ferguson MJ, Bahary JP, Schaeffer EM, Sandler HM, Tran PT, Rodgers JP, Esteva A, Yamashita R, Feng FY. Artificial Intelligence Predictive Model for Hormone Therapy Use in Prostate Cancer. NEJM Evid. 2023 Aug;2(8):EVIDoa2300023. doi: 10.1056/EVIDoa2300023. Epub 2023 Jun 29. PMID 38320143
- [Derived] Alexander GS, Krc RF, Assif JW, Sun K, Molitoris JK, Tran P, Rana Z, Bentzen SM, Mishra MV. Conditional Risks of Biochemical Failure and Prostate Cancer-Specific Death in Patients Undergoing External Beam Radiotherapy: A Secondary Analysis of 2 Randomized Clinical Trials. JAMA Netw Open. 2023 Sep 5;6(9):e2335069. doi: 10.1001/jamanetworkopen.2023.35069. PMID 37751207
- [Derived] Spratt DE, Liu VYT, Michalski J, Davicioni E, Berlin A, Simko JP, Efstathiou JA, Tran PT, Sandler HM, Hall WA, Thompson DJS, Parliament MB, Dayes IS, Correa RJM, Robertson JM, Gore EM, Doncals DE, Vigneault E, Souhami L, Karrison TG, Feng FY. Genomic Classifier Performance in Intermediate-Risk Prostate Cancer: Results From NRG Oncology/RTOG 0126 Randomized Phase 3 Trial. Int J Radiat Oncol Biol Phys. 2023 Oct 1;117(2):370-377. doi: 10.1016/j.ijrobp.2023.04.010. Epub 2023 May 2. PMID 37137444
- [Derived] Kim S, Kong JH, Lee Y, Lee JY, Kang TW, Kong TH, Kim MH, You SH. Dose-escalated radiotherapy for clinically localized and locally advanced prostate cancer. Cochrane Database Syst Rev. 2023 Mar 8;3(3):CD012817. doi: 10.1002/14651858.CD012817.pub2. PMID 36884035
- [Derived] Michalski JM, Moughan J, Purdy J, Bosch W, Bruner DW, Bahary JP, Lau H, Duclos M, Parliament M, Morton G, Hamstra D, Seider M, Lock MI, Patel M, Gay H, Vigneault E, Winter K, Sandler H. Effect of Standard vs Dose-Escalated Radiation Therapy for Patients With Intermediate-Risk Prostate Cancer: The NRG Oncology RTOG 0126 Randomized Clinical Trial. JAMA Oncol. 2018 Jun 14;4(6):e180039. doi: 10.1001/jamaoncol.2018.0039. Epub 2018 Jun 14. PMID 29543933
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 70.2 Gy | 79.2 Gy
Started | 769 | 763
Completed | 751 (Subjects with data available for the primary analysis are considered to have completed the study.) | 748 (Subjects with data available for the primary analysis are considered to have completed the study.)
Not Completed | 18 | 15
Not completed — Protocol Violation | 14 | 11
Not completed — Withdrawal by Subject | 4 | 4

BASELINE CHARACTERISTICS:
Population: All eligible patients who did not withdraw consent
Groups:
- Total: Total of all reporting groups
Arm/Group | 70.2 Gy | 79.2 Gy | Total
Number analyzed (Participants) | 751 | 748 | 1499
Age, Continuous [Median (Full Range); unit: years] | 71 [33 to 86] | 71 [49 to 87] | 71 [33 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 751 | 748 | 1499

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Survival time is defined as time from randomization to the date of death from any cause and is estimated by the Kaplan-Meier Method. Patients last know to be alive are censored at date of last contact.
Time Frame: From randomization to date of failure (death) or last follow-up. Analysis occurs after all patients have been potentially followed for 8 years.
Population: All eligible patients who did not withdraw consent
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 79.2 Gy: 79.2 Gy 3D-CRT/IMRT: Radiation will be delivered via 3D conformal radiation therapy (3D-CRT) or intensity modulated radiation therapy (IMRT) in 1.8 Gy minimum dose fractions to a total of 79.2 Gy in 44 fractions . All fields treated once daily, five fractions per week. No more than 2% of the planning target volume and none of the clinical target volume may receive less than 79.2 Gy.
Arm/Group | 70.2 Gy | 79.2 Gy
Number analyzed (Participants) | 751 | 748
percentage of participants | 88.5 [86.2 to 90.9] | 88.1 [85.7 to 90.4]
Statistical Analysis 1: Comparison: 70.2 Gy vs 79.2 Gy; The original target sample size was 1520 patients with a requirement of 715 deaths to test the hypothesis of overall survival (OS) efficacy of the 79.2 Gy arm. The trial was designed to detect a hazard ratio (HR) of 1.30 (standard/high-dose) with 90% statistical power at a one-sided significance level of 0.025; Test type: Superiority or Other; p = 0.98, Log Rank — Two-sided test, significance level = 0.05; Hazard Ratio (HR) = 1.0, 95% CI 2-sided [0.83 to 1.2] — Reference level = 70.2 Gy arm

2. Secondary Outcome: Prostate-specific Antigen (PSA) Failure by American Society for Therapeutic Radiology and Oncology (ASTRO) Definition
Description: Failure is defined as having 3 consecutive elevations of post-treatment PSA or starting hormones after one or more elevations in post-treatment PSA but before three consecutive elevations were documented. The failure day date was the midpoint between last non-rising PSA and first PSA rise. Failure rates are estimated by the cumulative incidence method. Patients last known to be alive are censored at date of last contact.
Time Frame: From randomization to date of failure (3 consecutive rises) or death or last follow-up. Analysis occurred after patients have been potentially followed for 5 years.
Population: All eligible patients who did not withdraw consent
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 70.2 Gy | 79.2 Gy
Number analyzed (Participants) | 751 | 748
percentage of participants | 40.2 [36.6 to 43.7] | 25.2 [22.1 to 28.4]
Statistical Analysis 1: Comparison: 70.2 Gy vs 79.2 Gy; Test type: Superiority or Other; p < 0.0001, Gray's test — Two-sided significance level = 0.05; Reference arm is 70.2 Gy arm; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.50 to 0.70]

3. Secondary Outcome: Disease Specific Survival
Description: Survival time is defined as time from randomization to the date of death due to prostate cancer and is estimated by the cumulative incidence method. Patients last know to be alive are censored at date of last contact. Death due to prostate cancer was defined as primary cause of death certified as due to prostate cancer, or death in association with any of the following conditions: Further clinical tumor progression occurring after initiation of salvage anti-tumor therapy, a rise (that exceeds 1.0 ng/ml) in the serum PSA level on at least two consecutive occasions that occurred during or after salvage androgen suppression therapy, or disease progression in the absence of any anti-tumor therapy.
Time Frame: From randomization to date of failure (death due to prostate cancer) or death from other cause or last follow-up. Analysis occurs at the same time as the primary endpoint.
Population: All eligible patients who did not withdraw consent
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 70.2 Gy | 79.2 Gy
Number analyzed (Participants) | 751 | 748
percentage of participants | 1.4 [0.7 to 2.5] | 0.8 [0.4 to 1.8]
Statistical Analysis 1: Comparison: 70.2 Gy vs 79.2 Gy; Test type: Superiority or Other; p = 0.14, Gray's test; Two-sided significance level = 0.05; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.38 to 1.15] — Reference level is 70.2 Gy arm

4. Secondary Outcome: Local Progression
Description: Failure time is defined as time from randomization to the date of progression (increase in palpable abnormality), failure of regression of the palpable tumor by two years, and redevelopment of a palpable abnormality after complete disappearance of previous abnormalities. Failure rates are estimated by the cumulative incidence method. Patients last know to be alive are censored at date of last contact.
Time Frame: From randomization to date of failure (local progression) or death or last follow-up. Analysis occurs at the same time as the primary endpoint.
Population: All eligible patients who have not withdrawn consent
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 70.2 Gy | 79.2 Gy
Number analyzed (Participants) | 751 | 748
percentage of participants | 3.5 [2.3 to 5] | 1.8 [1 to 3]
Statistical Analysis 1: Comparison: 70.2 Gy vs 79.2 Gy; Test type: Superiority or Other; p = 0.0001, Gray's test; Two-sided significance level = 0.05; Hazard Ratio (HR) = 0.41, 95% CI 2-sided [0.25 to 0.66] — Reference level = 70.2 Gy arm

5. Secondary Outcome: Distant Metastases
Description: Failure time is defined as time from randomization to the date of documented regional nodal recurrence or development of distant disease. Failure rates are estimated by the cumulative incidence method. Patients last know to be alive are censored at date of last contact.
Time Frame: From randomization to date of failure (distant metastasis) or death or last follow-up. Analysis occurs at the same time as the primary endpoint.
Population: All eligible patients who have not withdrawn consent
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 70.2 Gy | 79.2 Gy
Number analyzed (Participants) | 751 | 748
percentage of participants | 3.1 [2.0 to 4.6] | 2.2 [1.3 to 3.5]
Statistical Analysis 1: Comparison: 70.2 Gy vs 79.2 Gy; Test type: Superiority or Other; p = 0.051, Gray's test — Two-sided significance level = 0.05; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.42 to 1.01] — Reference level is the 70.2 Gy level

6. Secondary Outcome: Grade 2 or Greater Genitourinary or Gastrointestinal Toxicity
Description: Rate of acute 2+ grade genitourinary(GU)/gastrointestinal(GI) toxicity graded by Common Toxicity Criteria (CTC) version 2.0
Time Frame: From the start of treatment to 90 days. Analysis occurs at the same time as the primary endpoint
Population: Eligible patients with acute adverse event data who did not withdraw consent.
Measure: Number; unit: percentage of participants
Arm/Group | 70.2 Gy | 79.2 Gy
Number analyzed (Participants) | 733 | 728
percentage of participants | 18.8 | 21.0
Statistical Analysis 1: Comparison: 70.2 Gy vs 79.2 Gy; Test type: Superiority or Other; p = 0.29, Chi-squared — Two-sided significance level = 0.05

7. Secondary Outcome: Percentage of Participants With Erectile Disfuction at 12 Months
Description: The International Index of Erectile Function Questionnaire (IIEF) is the primary measure for erectile function (ED). IIEF question number 1 ("How often were you able to get an erection during sexual activity?") is scored from: none/almost never (response 0-1) or < half the time (response 2-3) to most times/almost always/always (response 4-5). A response of 0 to 3 on question number 1 of the IIEF is considered erectile dysfunction.
Time Frame: Twelve months from randomization
Population: Eligible patients with a response of 4 or 5 (most times/almost always/always) to IIEF question 1 at baseline
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 70.2 Gy | 79.2 Gy
Number analyzed (Participants) | 134 | 145
percentage of participants | 38.06 [29.84 to 46.28] | 49.66 [41.52 to 57.79]
Statistical Analysis 1: Comparison: 70.2 Gy vs 79.2 Gy; With an expected percentage of erectile disfunction (ED) at 12 months of 29%, a two-sided significance level of 0.05, and 688 patients per arm provides 90% statistical power to detect a reduction in ED to 19%. This calculation assumes 26% ED at baseline and 80% compliance at 12 months. Only participants with baseline ED are analyzed; Test type: Superiority; p = 0.0513, Chi-squared; Two-sided significance level = 0.05

8. Secondary Outcome: Number of Participants With Improved, Stable, and Declined Spitzer Quality of Life Index (SQLI) at 12 Months
Description: The SQLI measures quality of life for patients with cancer and other chronic diseases. Possible scores range from 0 to 10, with higher scores indicating a better outcome. Change from Baseline is defined as 12 month SQLI - baseline SQLI and is classified as follows:
  Improvement: when change >= to the standard error of measurement with reliability quotient of 0.5 (SEM); Stable: when -SEM < change < SEM; Declined: when change <= SEM.
Time Frame: Baseline and 12 months from randomization
Population: Eligible participants with baseline and 12 month SQLI
Measure: Count of Participants; unit: Participants
Arm/Group | 70.2 Gy | 79.2 Gy
Number analyzed (Participants) | 547 | 517
Participants
  Improved | 91 | 91
  Stable | 366 | 331
  Declined | 90 | 95
Statistical Analysis 1: Comparison: 70.2 Gy vs 79.2 Gy; Test type: Superiority; p = 0.59, Chi-squared; Two-sided significance level = 0.05

9. Secondary Outcome: Quality Adjusted Survival by SQLI
Time Frame: From randomization to 5 years.
Population: This analysis will not be done because we are unable to find the required algorithm for converting SQLI scores into utilities, which is needed for quality adjusted survival analysis.
Arm/Group | 70.2 Gy | 79.2 Gy
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Tumor Control Probability
Time Frame: From randomization to date of failure (tumor progression) or last follow-up. Analysis can occur any time after the primary endpoint analysis.
Reporting Status: Not Posted, anticipated posting 2023-12

11. Secondary Outcome: Normal Tissue Complication Probability
Time Frame: From randomization to last follow-up. Analysis can occur any time after the primary endpoint analysis.
Reporting Status: Not Posted, anticipated posting 2023-12

ADVERSE EVENTS:
Description: Eligible patients with toxicity data who did not withdraw consent. Subjects experiencing more than one of a given adverse event are counted only once for that adverse event.
Groups:
- 70.2 Gy: 70.2 Gy 3D-CRT/IMRT: Radiation will be delivered via 3D conformal radiation therapy (3D-CRT) or intensity modulated radiation therapy (IMRT) in 1.8 Gy minimum dose fractions to a total of 70.2 Gy in 39 Fractions . All fields treated once daily, five fractions per week. No more than 2% of the planning target volume and none of the clinical target volume may receive less than 70.2 Gy.
- 79.2 Gy: 79.2 Gy 3D-CRT/IMRT: Radiation will be delivered via 3D conformal radiation therapy (3D-CRT) or intensity modulated radiation therapy (IMRT) in 1.8 Gy minimum dose fractions to a total of 70.2 Gy in 44 Fractions . All fields treated once daily, five fractions per week. No more than 2% of the planning target volume and none of the clinical target volume may receive less than 79.2 Gy.
Arm/Group | 70.2 Gy | 79.2 Gy
Serious Adverse Events (participants affected / at risk) | 30/744 | 43/737
Other Adverse Events (participants affected / at risk) | 714/744 | 704/737
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 70.2 Gy (N=744) | 79.2 Gy (N=737)
Left ventricular failure (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 2 | 1
Abdominal pain NOS (Gastrointestinal disorders) | 1 | 0
Diarrhea (with colostomy) (Gastrointestinal disorders) | 0 | 1
Diarrhea NOS (Gastrointestinal disorders) | 2 | 0
Late RT Toxicity: Bowel : NOS (Gastrointestinal disorders) | 1 | 1
Late RT Toxicity: Other GI : NOS (Gastrointestinal disorders) | 1 | 4
Chest pain (General disorders) | 1 | 0
Injection site reaction NOS (General disorders) | 0 | 1
Late RT Toxicity: Other : NOS (General disorders) | 1 | 3
Pain due to radiation (General disorders) | 0 | 2
Pain-other (General disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 2
Late RT Toxicity: Bladder/Other GU: NOS (Renal and urinary disorders) | 0 | 3
Urinary incontinence (Renal and urinary disorders) | 21 | 21
Urinary retention (Renal and urinary disorders) | 1 | 2
Dyspnea NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin-Other (Skin and subcutaneous tissue disorders) | 0 | 2
Hemorrhage-Other (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 70.2 Gy (N=744) | 79.2 Gy (N=737)
Diarrhea NOS (Gastrointestinal disorders) | 58 | 50
Late RT Toxicity: Bowel : NOS (Gastrointestinal disorders) | 90 | 128
Late RT Toxicity: Other GI : NOS (Gastrointestinal disorders) | 90 | 107
Proctitis NOS (Gastrointestinal disorders) | 33 | 45
Fatigue (General disorders) | 51 | 51
Late RT Toxicity: Other : NOS (General disorders) | 68 | 90
Dysuria (Renal and urinary disorders) | 52 | 53
Late RT Toxicity: Bladder/Other GU: NOS (Renal and urinary disorders) | 99 | 126
Urinary frequency (Renal and urinary disorders) | 566 | 585
Urinary incontinence (Renal and urinary disorders) | 234 | 229
Impotence (Reproductive system and breast disorders) | 611 | 599

LIMITATIONS AND CAVEATS:
The data monitoring committee (DMC) recommended early reporting of the trial when the third interim analysis futility boundary was crossed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.